CLINICAL TRIAL: NCT05288985
Title: Prospective, Randomised, Controlled Pilot Study Evaluating the Impact of Loco-regional Analgesia Following Placement of Erector Spinae Plane Catheter in Addition to Systemic Analgesia in Patients With Thoracic Trauma
Brief Title: Impact of Loco-regional Analgesia Following Placement of Erector Spinae Plane Catheter in Addition to Systemic Analgesia in Patients With Thoracic Trauma
Acronym: ERECTRAUTHO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHD21_0043
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-07

CONDITIONS: Trauma Abdomen
MeSH Terms: conditions — Abdominal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane catheter group in addition to Systemic Analgesia (Experimental)
  Interventions: Device: Erector spinae plane catheter group in addition to Systemic Analgesia
- Systemic Analgesia Only Group (Active Comparator)
  Interventions: Drug: Systemic Analgesia Only Group

INTERVENTIONS:
Device: Erector spinae plane catheter group in addition to Systemic Analgesia — Erector spinae plane catheter is placed in the post-interventional surveillance room in the operating theatre by an anaesthetist-intensive care physician or in the MIR department by the intensive care physician in charge of the patient within 2 hours after randomisation. The local anaesthetic injected into the catheter is Ropivacaine, prescribed according to a protocol of continuous flow, bolus and refractory period. The catheter is repositioned if a secondary displacement occurs.
  Arms: Erector spinae plane catheter group in addition to Systemic Analgesia
Drug: Systemic Analgesia Only Group — Systemic analgesia alone consists only of the 3 levels of analgesic treatment
  Arms: Systemic Analgesia Only Group

SUMMARY:
The management of analgesia is the key issue in the management of a thoracic trauma patient to prevent respiratory complications.

A multimodal approach is recommended but the question of the most suitable loco-regional analgesia technique remains. It must combine effectiveness and simplicity with the least risk to the patient. Today, epidural analgesia is the technique of choice, but it has certain disadvantages: difficulties in performing it at the thoracic level, undesirable effects, complications, and numerous contraindications.

The investigator propose to carry out a single-centre, prospective, randomised, controlled pilot study evaluating the impact of loco-regional analgesia following the placement of erector spinae plane catheter in addition to systemic analgesia in patients with unilateral thoracic trauma.

The aim is to demonstrate the effectiveness of this technique, which has fewer disadvantages than epidural analgesia. The interest of this study is thus to decrease the respiratory morbidity of thoracic trauma patients by avoiding a maximum of complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Unibilateral chest trauma with fracture > 2 ribs on one side
* Admission to Intensive Care Medicine
* Non-intubated patient, able to respond to a pain scale score and perform a vital capacity
* Numerical Scale > 3 on forced inspiration despite use of systemic analgesics
* CV ≤ 80% theoretical at inclusion
* Time < 24 hours from admission to the service to inclusion
* Time < 48h between trauma and inclusion
* Patient affiliated to the social security system or entitled to it
* Patient able to understand the protocol, having agreed to participate in the study and having given express oral consent

Exclusion Criteria:

* Intubated, ventilated patient
* Indication for laparotomy or thoracotomy
* Spinal cord injury
* Severe head injury
* Bilateral thoracic trauma
* Patient included in a category 1 clinical interventional study involving analgesic treatment
* Patients under legal protection or deprived of liberty
* Pregnant or breastfeeding women, or women with childbearing potential without effective contraception
* Refusal to participate
* Unable to understand the protocol and its requirements and/or unable to give express oral consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2026-01-14 (Estimated); Study Completion 2026-01-14 (Estimated)

PRIMARY OUTCOMES:
Change in vital capacity between inclusion and 24 hours after inclusion. | Inclusion and 24 hours after inclusion
  Vital capacity is the maximum amount of air that can be breathed in and out of the lungs in one breath. It is therefore a reflection of the thoracic expansion capacity. It is expressed as a percentage of the theoretical or predicted value, which is calculated from the patient's age, height, sex and ethnic group. It is measured with the CareFusion spirometer of the MIR department, inspiration must be maximal and expiration must last at least 6 seconds in theory (3 seconds tolerated by the spirometer). 2 measurements are made and the best of the 2 is chosen.

CONTACTS AND LOCATIONS:
Overall Officials: Laureen GUILLEMIN, Principal Investigator — Centre Hospitalier Départemental Vendée
Locations (1):
- Centre Hospitalier Départemental Vendée, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No